CLINICAL TRIAL: NCT03460717
Title: Peripheral Nerve Field Stimulation by Thermal Micro-cautery for Painful Knee Osteoarthritis: Non Randomised Controlled Trial
Brief Title: Thermal Micro-cautery for Painful Knee Osteoarthritis
Acronym: TMC-PKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Children's Hospital, Tallaght (Other)
Responsible Party: Principal Investigator, Camillus Power, Director of Pain Medicine, The National Children's Hospital, Tallaght
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-10 Chairman's Action (3)
Record Dates: First submitted 2018-02-09; First posted 2018-03-09 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2018-03

CONDITIONS: Chronic Pain Syndrome

STUDY DESIGN:
Intervention Model Description: intervention offered and those who decline are followed as a waiting list control
Who Masked: Investigator, Outcomes Assessor
Masking Description: the person performing the intervention and the assessment are different
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: PNFS-TMC (Experimental): Procedure- The patients in the intervention group were examined and the most painful points over the knee with the avoidance of the proposed site for skin incision for a future knee replacement operation were marked. The marked points received an intervention in the form of application of Peripheral Nerve Field Stimulation by Thermal Micro-Cautery (PNFS-TMC), an intense heat by metal rod was applied to the painful points for 0.3 to 0.5 seconds. The patients to receive 4 sessions over a period of 8 weeks with 2 weeks rest after every session.
  Interventions: Other: Peripheral Nerve Field Stimulation by Thermal Micro-Cautery
- Control group: Stepladder analgesics (No Intervention): Patients with painful knee osteoarthritis and on the waiting list for a total knee replacement surgery and declined to have PNFS-TMC were included in the control group. The control group received the stepladder analgesic protocol for pain management. The analgesic protocol was managed by the orthopaedic team without any interference by the investigators.

INTERVENTIONS:
Other: Peripheral Nerve Field Stimulation by Thermal Micro-Cautery — The most painful points over the knee received an intense heat by a metal rod for 0.5 seconds.
  Arms: Intervention group: PNFS-TMC

SUMMARY:
To trial a traditional pain management technique from Ayurveda in a modern way - the technique involves micro - cautery to painful areas in knee osteoarthritis for patients on a waiting list for knee replacement. The Investigators will include a waiting list control series.

DETAILED DESCRIPTION:
The Research and Ethics Committee at Tallaght University Hospital approved the recruitment of patient into the study by invitation. Patients who accepted the invitation were enrolled into the intervention group and patients who declined the invitation were enrolled into the control group and both groups were followed up for 8 week period. Agnikarma is a traditional surgical technique (thermal cautery) described in ancient surgical manuscripts for the treatment of severe persistent pain.

It applies intense heat to points of maximum pain agreed with the patient pre procedure. The heat is applied by a metal rod (Shalaka) heated in an open naked flame. The rod is applied to the skin at the agreed pain point in an even manner and generates a micro second degree burn. A traditional herbal cream is then applied which cools the application as reported by the patient. It is usual to allow skin healing to occur before the application of further heat (1-2 weeks). The pain points can move within a painful area and the technique best works with precise application to the current pain point. So before each application the precise points are agreed with the patient in advance by demarcating the painful area with a pen and searching for the points of maximum tenderness within that field.

The purpose of this study was simply to define if indeed this technique delivers pain relief as observed in practice. The investigators chose one group to study - painful knee arthritis. In this condition patients often wait many years for the definitive procedure and run some risks with current pain relief treatment. As these patients were not the normal attendees at a pain clinic the investigators decided in advance to limit the study to 4 applications over a 4- 8 week period, the latter to allow for different speeds at which the skin might heal. The investigators recruited both our interventional group and waiting list control group from the same orthopedic waiting list.

ELIGIBILITY:
Inclusion Criteria:

* awaiting knee replacement surgery on an orthopaedic waiting list

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change in VAS score reduction after 4 sessions | VAS score was recorded every two weeks, after each session with a total of 4 sessions over 8 weeks. 2 weeks interval between sessions
  To measure the change in a visual analogue scale is a numerical ruler of 10 cm in length with each centimetre marked and the patient chooses a number between one and ten to score their pain where zero is no pain and 10 is the worst pain that the subject can imagine.

SECONDARY OUTCOMES:
Change in activity levels | The objective activity score was recorded every two weeks after each session with a total of 4 sessions over 8 weeks
  The change in the activity subjective scores reported by the patient as follow; score 1 means improved , score 2 means worse and score 3 means no change
Change in sleep pattern | The change in the sleep pattern was recorded every two weeks after each session with a total of 4 sessions over 8 weeks
  The change in the subjective scores reported by patient as follows, score 1 means improved, 2 means worse and 3 means the same as before
Change in medication use | The change in the medication use was recorded every two weeks after each session with a total of 4 sessions over 8 weeks
  1 means improved as in less use of medication, 2 means worse more use of medication and 3 means the same use of analgesic medication

CONTACTS AND LOCATIONS:
Overall Officials: camillus power, MD, Principal Investigator — Tallaght University Hospital
Locations (1):
- Tallaght University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No